CLINICAL TRIAL: NCT05172245
Title: Phase 1/1b Study of AKT Inhibitor Ipatasertib With Chemoradiation for Locally Advanced Head and Neck Cancer
Brief Title: Testing the Addition of Ipatasertib to Usual Chemotherapy and Radiation for Head and Neck Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-13901; NCI-2021-13901 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 032204; 10492 (Other: University Health Network Princess Margaret Cancer Center LAO); 10492 (Other: CTEP); UM1CA186644 (NIH)
Record Dates: First submitted 2021-12-28; First posted 2021-12-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Clinical Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Head and Neck Carcinoma of Unknown Primary; Locally Advanced Head and Neck Squamous Cell Carcinoma; Locally Advanced Hypopharyngeal Squamous Cell Carcinoma; Locally Advanced Laryngeal Squamous Cell Carcinoma; Locally Advanced Nasal Cavity Squamous Cell Carcinoma; Locally Advanced Oral Cavity Squamous Cell Carcinoma; Locally Advanced Oropharyngeal Squamous Cell Carcinoma; Locally Advanced Paranasal Sinus Squamous Cell Carcinoma; Locally Advanced Sinonasal Squamous Cell Carcinoma; Maxillary Sinus Squamous Cell Carcinoma; Stage III Hypopharyngeal Carcinoma AJCC v8; Stage III Laryngeal Cancer AJCC v8; Stage III Lip and Oral Cavity Cancer AJCC v8; Stage III Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage III Sinonasal Cancer AJCC v8; Stage IVA Hypopharyngeal Carcinoma AJCC v8; Stage IVA Laryngeal Cancer AJCC v8; Stage IVA Lip and Oral Cavity Cancer AJCC v8; Stage IVA Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVA Sinonasal Cancer AJCC v8; Stage IVB Hypopharyngeal Carcinoma AJCC v8; Stage IVB Laryngeal Cancer AJCC v8; Stage IVB Lip and Oral Cavity Cancer AJCC v8; Stage IVB Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVB Sinonasal Cancer AJCC v8
MeSH Terms: conditions — Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Carcinoma | interventions — Biopsy; Specimen Handling; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; ipatasertib; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation (ipatasertib, cisplatin, radiation therapy) (Experimental): Patients receive ipatasertib PO QD or Monday, Wednesday, and Friday depending on dose level on days 1-28 of each cycle. Patients also receive cisplatin IV weekly on day 1 of cycle 1, weeks 1-4 and day 1 of cycle 2, weeks 1-3 for 7 doses. Patients undergo RT daily (Monday-Friday) for 35 fractions during weeks 1-7. Treatment repeats every 28 days for a total of 2 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo PET/CT, CT, or MRI during screening, follow-up, and as clinically indicated. Patients undergo blood sample collection on trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Ipatasertib; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy
- Dose Expansion (ipatasertib, cisplatin, radiation therapy) (Experimental): Patients receive ipatasertib PO MTD on days 2-28 or 3-28 of cycle 1 and 1-28 of subsequent cycles. Patients also receive cisplatin IV weekly on day 1 of cycle 1, weeks 1-4 and day 1 of cycle 2, weeks 1-3 for 7 doses. Patients undergo RT daily (Monday-Friday) for 35 fractions during weeks 1-7. Treatment repeats every 28 days for a total of 2 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo PET/CT, CT, or MRI during screening, follow-up, and as clinically indicated. Patients undergo blood sample collection and tumor biopsy on trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Ipatasertib; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
  Arms: Dose Expansion (ipatasertib, cisplatin, radiation therapy)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Ipatasertib — Given PO
  Other Names: GDC 0068; GDC-0068; GDC0068; RG 7440; RG-7440; RG7440
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase I/Ib trial tests the safety and best dose of ipatasertib in combination with the usual treatment approach using chemotherapy together with radiation therapy ("chemo-radiation") in patients with head and neck cancer. Ipatasertib is in a class of medications called protein kinase B (AKT) inhibitors. It may stop the growth of tumor cells and may kill them. Cisplatin, which is a chemotherapy used in this trial, is in a class of medications known as platinum-containing compounds. It works by killing, stopping or slowing the growth of cancer cells. Radiation therapy uses high energy to kill tumor cells and shrink tumors. Giving ipatasertib in combination with chemo-radiation may be better than chemo-radiation alone in treating patients with advanced head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of ipatasertib in combination with definitive chemoradiation in locally advanced head and neck squamous cell carcinoma (HNSCC) based on dose-limiting toxicities (DLTs).

SECONDARY OBJECTIVES:

I. To assess acute and late toxicities, based on Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

II. To assess long-term swallowing function, based on gastric tube dependency at 6 and 12 months that is different from baseline.

III. To determine duration and completion rate of prescribed radiation and chemotherapy.

IV. To determine pharmacokinetic profile of ipatasertib in combination with cisplatin and radiation therapy, based on peak and trough blood levels in patients administered ipatasertib orally.

V. To determine pharmacodynamic effects of ipatasertib at the MTD, based on pAKT, pS6 and pPRAS40 as markers of AKT pathway inhibition, and gamma-H2AX as a marker of radiosensitization.

VI. To observe and record anti-tumor activity (objective response rate by Response Evaluation Criteria in Solid Tumors [RECIST] criteria, locoregional control, relapse-free survival, and overall survival) of the combination of ipatasertib, cisplatin, and radiation therapy in patients with HNSCC.

VII. To correlate efficacy outcomes with tumor genotype, based on whole exome sequencing of pre-treatment biopsy specimens.

OUTLINE: This is a phase I, dose-escalation study of ipatasertib in combination with fixed-dose cisplatin and radiation therapy followed by a dose-expansion study.

DOSE ESCALATION:

Patients receive ipatasertib orally (PO) once daily (QD) or Monday, Wednesday, and Friday depending on dose level on days 1-28 of each cycle. Patients also receive cisplatin intravenously (IV) weekly on day 1 of cycle 1, weeks 1-4 and day 1 of cycle 2, weeks 1-3 for 7 doses. Patients undergo radiation therapy (RT) daily (Monday-Friday) for 35 fractions during weeks 1-7. Treatment repeats every 28 days for a total of 2 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo positron emission tomography (PET)/computed tomography (CT), CT, or magnetic resonance imaging (MRI) during screening, follow-up, and as clinically indicated. Patients undergo blood sample collection on trial.

DOSE EXPANSION:

Patients receive ipatasertib PO MTD on days 2-28 or 3-28 of cycle 1 and 1-28 of subsequent cycles. Patients also receive cisplatin IV weekly on day 1 of cycle 1, weeks 1-4 and day 1 of cycle 2, weeks 1-3 for 7 doses. Patients undergo RT daily (Monday-Friday) for 35 fractions during weeks 1-7. Treatment repeats every 28 days for a total of 2 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo PET/CT, CT, or MRI during screening, follow-up, and as clinically indicated. Patients undergo blood sample collection and tumor biopsy on trial.

After completion of study treatment, patients are followed for 30 days and then every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed HNSCC (including tumors of the oropharynx, hypopharynx, larynx, oral cavity, nasal cavity, maxillary and other paranasal sinuses, and unknown primary of the head and neck), with measurable disease as per RECIST 1.1
* Oropharyngeal and unknown primary squamous cell cancers must test for human papilloma virus (HPV), for example by p16 immunohistochemistry (IHC), in situ hybridization (ISH), or polymerase chain reaction (PCR). HPV testing is not required for other HNSCC primary tumor sites

  * Patients with p16-positive tumors are eligible if clinical stage III (cT4 or cN3, M0) according to the American Joint Committee on Cancer (AJCC)/TNM Staging System, 8th edition (Ed.)
  * Patients with p16-negative (or not tested) tumors are eligible if clinical stage III-IVB (locally advanced but non-metastatic) according to the AJCC/TNM Staging System, 8th Ed.
* Must be candidate for concurrent, definitive cisplatin and radiation therapy as judged by the treating physician
* Able to swallow tablets at the time of enrollment
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of ipatasertib in combination with chemoradiation in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Life expectancy of greater than 3 months
* Absolute neutrophil count >= 3000/mcL
* Hemoglobin >= 10 g/dL
* Platelets >= 150,000/mcL
* Serum albumin >= 3 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN / 2 x institutional ULN
* Alkaline phosphatase (ALP) =< 2.0 x institutional ULN
* Partial thromboplastin time (PTT) (or activated [a]PTT) and international normalized ratio (INR) =< 1.5 institutional ULN (except for patients receiving anticoagulation therapy)
* Creatinine clearance (CLcr) > 60 mL/min

  * For this calculation, use the Cockroft-Gault formula
* Fasting glucose =< 150 mg/dL (8.3 mmol/L) and (when indicated) glycosylated hemoglobin (HbA1c ) =< 7.5% (58 mmol/mol)
* Human immunodeficiency virus (HIV)-infected patients are eligible if on effective anti-retroviral therapy with undetectable viral load within 6 months
* Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative hepatitis B virus surface antigen [HBsAg] test and a positive hepatitis B core antibody [HBcAb] test, accompanied by a negative HBV deoxyribonucleic acid [DNA] test) are eligible. Patients with chronic HBV infection are eligible if the HBV viral load is undetectable on suppressive therapy, if indicated. Patients undergoing current treatment with anti-viral therapy for HBV are ineligible
* Patients with a history of hepatitis C virus (HCV) infection are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA). Patients with HCV infection who are currently on treatment are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* The effects of ipatasertib on the developing human fetus are unknown. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for at least 28 days after the last dose of ipatasertib and agreement to refrain from donating eggs during this same period. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm during the treatment period and for 28 days after the last dose of ipatasertib
* Ability to understand and the willingness to sign a written informed consent document
* For the expansion cohort only, patients must agree to undergo mandatory on-treatment biopsies, and have tumors amenable to on-treatment biopsies. This is not applicable to the dose escalation cohort where no on-treatment biopsies are obtained

Exclusion Criteria:

* Primary tumor of nasopharynx, salivary, thyroid or parathyroid glands, or skin
* Distant metastases from the current HNSCC
* Prior treatment (e.g., chemotherapy, radiation, or definitive surgery) for the current locally advanced HNSCC is not permitted. Biopsies, including those performed under anesthesia, are not considered surgery. Patients who underwent prior definitive surgery alone for an early stage (T1-2N0) HNSCC which has now recurred with stage III-IVB disease at least 3 months after the initial surgery are eligible
* For patients with a prior history of another malignancy, no prior chemotherapy or radiation may have been administered within 6 weeks prior to study entry. Among patients who received prior radiation to the head and neck or adjacent anatomical site for another malignancy, there may be no overlap with current area to be irradiated
* Current use of any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ipatasertib or other agents used in study
* Treatment with strong inhibitors or inducers of CYP3A4 or P-glycoprotein within 2 weeks or 5 drug-elimination half-lives, whichever is longer, prior to initiation of study drug. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with uncontrolled intercurrent illness, including active infection
* Pregnant women are excluded from this study because ipatasertib is an oral AKT inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ipatasertib, breastfeeding should be discontinued if the mother is treated with ipatasertib. These potential risks may also apply to other agents used in this study
* Patients with type I or type II diabetes mellitus requiring insulin at study entry. Patients with non-insulin dependent type II diabetes mellitus are eligible, as are patients who are on a stable dose of oral diabetes medication >= 4 weeks prior to initiation of study treatment. Patients with a history of diabetes mellitus, an abnormal fasting glucose level, or other signs or symptoms indicating diabetes mellitus, must meet the laboratory eligibility criteria for fasting blood glucose and hemoglobin A1c
* History of or active inflammatory bowel disease (e.g., Crohn's disease and ulcerative colitis) or active bowel inflammation (e.g., diverticulitis)
* History of malabsorption syndrome or other condition that would interfere with enteral absorption or results in the inability or unwillingness to swallow pills
* Lung disease: pneumonitis, interstitial lung disease, idiopathic pulmonary fibrosis, cystic fibrosis, aspergillosis, active tuberculosis, or history of opportunistic infections (pneumocystis pneumonia or cytomegalovirus pneumonia)
* Known clinically significant history of liver disease consistent with Child Pugh Class B or C, including active viral or other hepatitis (e.g., positive for hepatitis B surface antigen [HBsAg] or hepatitis C virus [HCV] antibody at screening), or cirrhosis
* Grade >= 2 uncontrolled or untreated hypercholesterolemia (cholesterol > 300 mg/dL or > 7.75 mmol/L) or hypertriglyceridemia (triglycerides > 300 mg/dL or > 3.42 mmol/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and recommended phase 2 dose of ipatasertib in combination with definitive chemo-radiation | At the completion of dose escalation phase, up to 56 days from treatment start date
  Patients who receive at least 70% of the prescribed course of ipatasertib on radiation days will be evaluable for dose limiting toxicity assessment. After the escalation phase of the trial is completed, the MTD will be selected using the pooled-adjacent-violators algorithm, a type of isotonic regression, as specified in Liu and Yuan (2015).

SECONDARY OUTCOMES:
Acute and late toxicities | From 90 days after the end of radiation treatment up to 1 year from treatment completion date
  Will be assessed according to Common Terminology Criteria for Adverse Events version 5.0. Toxicities occurring > 90 days from the end of radiation will be considered late toxicities. This will include assessment of long-term swallowing function, based on gastric tube dependency at 6 and 12 months as compared to baseline due to the effects of the primary tumor. Descriptive statistics will be used to summarize these toxicities.
Duration and completion rate of prescribed radiation and chemotherapy | Up to 2 years
  Descriptive statistics will also be used to summarize the duration and completion rate of prescribed radiation and chemotherapy.
Objective response rate | Up to 2 years
  Assessed based on Response Evaluation Criteria in Solid Tumors, as well as locoregional control, relapse-free survival, and overall survival. Two-sample t-test, Mann-Whitney U test, or log rank test will be used where appropriate to analyze the correlation between efficacy outcomes and pre-treatment genotypic abnormalities in the AKT pathway based on whole exome sequencing and PTEN immunohistochemistry (IHC).
Pharmacokinetic (PK) profile of ipatasertib in combination with cisplatin | Up to 2 years
  Will be assessed using peak and trough blood levels in patients administered ipatasertib orally during weeks 2 and 3 of study treatment. The combined therapy will be compared to historical PK data for drug alone, in order to assess for a drug-drug interaction.
Pharmacodynamic effects of ipatasertib | Up to 2 years
  Based on pAKT, pS6 and PRAS40 as markers of AKT pathway inhibition, and gamma-H2AX as a marker of radiosensitization. Two-sample t-test and Mann-Whitney U test will be used where appropriate to compare values before and after the addition of ipatasertib to chemoradiation.
Locoregional control | From start of treatment to cancer recurrence at the site of the primary tumor or the regional lymph nodes, assessed up to 2 years
  Two-sample t-test, Mann-Whitney U test, or log rank test will be used where appropriate to analyze the correlation between efficacy outcomes and pre-treatment genotypic abnormalities in the AKT pathway based on whole exome sequencing and PTEN IHC.
Relapse-free survival | From start of treatment to the time of cancer recurrence or death, whichever occurs first, assessed up to 2 years
  Two-sample t-test, Mann-Whitney U test, or log rank test will be used where appropriate to analyze the correlation between efficacy outcomes and pre-treatment genotypic abnormalities in the AKT pathway based on whole exome sequencing and PTEN IHC.
Overall survival | From the start of treatment that patients are still alive, assessed up to 2 years
  Two-sample t-test, Mann-Whitney U test, or log rank test will be used where appropriate to analyze the correlation between efficacy outcomes and pre-treatment genotypic abnormalities in the AKT pathway based on whole exome sequencing and PTEN IHC.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm D Mattes, Principal Investigator — University Health Network Princess Margaret Cancer Center LAO
Locations (18):
- United States (17):
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm